CLINICAL TRIAL: NCT01453491
Title: A Phase 1b, Exploratory Study to Assess the Safety, Tolerability, Colonic Tissue Exposure, and Anti-Inflammatory Effects of Two Different Doses of SRT2104 in Subjects With Mild to Moderate Ulcerative Colitis
Brief Title: A Phase 1b Study to Assess the Safety and Anti-inflammatory Effects of Two Different Doses of SRT2104 in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirtris, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 115951
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — SRT2104

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50mg SRT2104 (Experimental): Single oral administration of 50mg SRT2104 study drug will be supplied as 25 mg and 250 mg capsules and will be taken orally once daily for 56 days. SRT2104 is to be taken at approximately the same time every morning, in the fasted state. Water is permitted ad libitum. Subjects are allowed to consume liquids but should refrain from eating solid food for approximately 1 hour after dosing.
  Interventions: Drug: SRT2104
- 500mg SRT2104 (Experimental): Single oral administration of 500mg SRT2104 will be taken orally once daily for 56 days. SRT2104 is to be taken at approximately the same time every morning, in the fasted state. Water is permitted ad libitum. Subjects are allowed to consume liquids but should refrain from eating solid food for approximately 1 hour after dosing.
  Interventions: Drug: SRT2104

INTERVENTIONS:
Drug: SRT2104 — SRT2104 drug substance is a new chemical entity which is supplied as a fine, yellowish/amber powder. The SRT2104 investigational product is prepared by packing 25mg or 250 mg of micronized SRT2104 powder with no additional additives into a size 00 opaque, hard gelatin capsule. All subjects will be provided with one dosing bottle per day that contains two 25 mg or 250 mg SRT2104 capsules for oral ingestion.

SUMMARY:
The purpose of this research study is to:

* 1) Test the safety and tolerability of 2 different oral doses of SRT2104 in subjects with ulcerative colitis
* 2) Determine the amount of SRT2104 measured from a single blood sample in addition to colon and/or rectal tissue samples (biopsies)
* 3) Determine whether SRT2104 has any anti-inflammatory effect on the colon and/or rectum when taken orally for 8 weeks
* 4) Determine whether SRT2104 causes any detectable changes to specific biomarkers. A biomarker is a biological marker (or substance such as a protein) that is used as an indicator of changes in a biological state that corresponds to the risk or progression of a disease.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderately active ulcerative colitis as evidenced by Mayo score 6-10 (inclusive) with rectal bleeding score ≥1, endoscopy score between 2-3 (inclusive), and physician's rating of disease activity <3 at Day -5
* Colonic inflammation extending proximal to the rectum (i.e., greater than 15 cm in extent) on baseline sigmoidoscopy at Day -5
* Confirmed diagnosis of ulcerative colitis for at least 3 months prior to the Screening Visit (Visit 1)
* Male or female between 18 and 75 years, inclusive
* Body weight >50 kg and BMI ≥18 kg/m^2 at Screening (Visit 1)
* Capable of giving written informed consent, and willing and able to comply with the requirements of the protocol
* Female subjects of child-bearing potential must be willing to use reliable contraception from Visit 1 through the follow-up visit (Day 70)

Exclusion Criteria:

* Suspicion of Crohn's disease, indeterminate colitis, microscopic colitis, segmental colitis associated with diverticulosis, ischemic colitis, or radiation-induced colitis based on medical history, endoscopy, and/or histological findings
* Presence of infectious colitis as evidenced by positive stool culture for enteric pathogens or positive stool Clostridium difficile cytotoxin assay at Visit 1
* Presence of chronic liver disease, with the exception of known Gilbert's syndrome
* A positive pre-study Hepatitis B surface antigen, Hepatitis C antibody or HIV at Visit 1
* Past or present disease that is judged by the investigator to have the potential to interfere with the study procedures or compromise the subject's safety
* History of malignant neoplasm within the past 5 years, other than localized basal cell carcinoma, squamous cell carcinoma, or carcinoma in situ that has been resected or definitively treated with standard approaches
* Prior diagnosis of flat colonic dysplasia or unresected raised colonic dysplasia (adenoma-like lesion or mass)
* History of regular alcohol consumption within 6 months of the Screening (Visit 1) defined as an average weekly intake of >14 drinks (one drink is defined as 12 ounces of beer, 5 ounces of wine, or 1.5 ounces of 80 proof distilled spirits) or presence of recreational drug abuse or dependence
* Known bleeding disorders
* Bowel surgery within 12 months prior to Visit 1
* History of colectomy or partial colectomy
* Treatment with oral aminosalicylates at doses >4.8 g per day or aminosalicylate dose modification (except transient shift lasting up to 3 days) within 4 weeks prior to study Day -5 (Note: if on this type of treatment, the dose must remain constant throughout the study treatment period)
* Treatment with rectal aminosalicylates at any dose within 2 weeks of study Day -5
* Treatment with systemic or rectal corticosteroids within 4 weeks of study Day -5
* Treatment with TNFα inhibitors or other biologics within 2 months prior to study Day -5
* Treatment with other immunosuppressants (azathioprine or 6-mercaptopurine), if initiated within 3 months prior to study Day -5, or if changed in terms of dose within 3 months prior to study Day -5 (Note: if on this type of treatment, the dose must remain constant throughout the study treatment period)
* Regular use of pro-biotic or prebiotic preparations within 4 weeks of study Day -5 visit
* Regular use of non-steroidal anti-inflammatories (NSAIDS) or aspirin, except low dose (cardioprotective ≤325 mg/day) aspirin, within 7 days prior to study Day -5
* Participation in a clinical trial and treatment with an study drug within 3 months prior to Visit 1
* Have a clinically significant finding on a chest X-ray performed at Visit 1 or within 3 months of Visit 1
* Have an abnormal 12-lead electrocardiogram (ECG) with one or more changes considered to be clinically significant on medical review
* Renal or liver impairment based on laboratory values obtained at Visit 1 and defined as:

  * serum creatinine level of ≥1.4 mg/dL for females and ≥1.5 mg/dL for males, or
  * AST and/or ALT ≥2x upper limit of normal (ULN), or
  * bilirubin > 1.5xULN (an isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin is <35%)
  * Hemoglobin less than 8.5 g/dL at Visit 1
  * Have any other reason which, in the opinion of the investigator, would confound the conduct or interpretation of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-02-13 (Actual); Primary Completion 2013-03-18 (Actual); Study Completion 2013-03-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and incidence of adverse events will be used as a measure of safety and tolerability of 50 mg and 500 mg of SRT2104 after repeat dosing for up to eight weeks in subjects with mild to moderate ulcerative colitis | 75 days
SRT2104 concentration in colonic tissue will be measured via endoscopic biopsy after repeat dosing for up to 8 weeks in subjects with mild to moderate ulcerative colitis | 56 days

SECONDARY OUTCOMES:
Endoscopic scoring of colonic lesions assessed during flexible sigmoidoscopy will be used as a measure of the anti-inflammatory effect of SRT2104 after 8 weeks of treatment in subjects with mild to moderate ulcerative colitis | 75 days
Mayo score and Partial Mayo score will be used as a measure of the anti-inflammatory effect of SRT2104 after 8 weeks of treatment in subjects with mild to moderate ulcerative colitis | 75 days
Simple Clinical Colitis Activity Index (SCCAI) will be used as a measure of the anti-inflammatory effect of SRT2104 after 8 weeks of treatment in subjects with mild to moderate ulcerative colitis | 75 days
Fecal calprotectin will be used as a measure of the anti-inflammatory effect of SRT2104 after 8 weeks of treatment in subjects with mild to moderate ulcerative colitis | 75 days
Histopathologic scoring of colonic tissue biopsies obtained via flexible sigmoidoscopy will be used as a measure of the anti-inflammatory effect of SRT2104 after 8 weeks of treatment in subjects with mild to moderate ulcerative colitis | 75 days
SRT2104 concentration in plasma will be measured after repeat dosing for up to 8 weeks in subjects with mild to moderate ulcerative colitis | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (13):
- United States (13):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Bristol, Connecticut
  - GSK Investigational Site, Owensboro, Kentucky
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Chesterfield, Michigan
  - GSK Investigational Site, Great Neck, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Beavercreek, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Jackson, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Sands BE, Joshi S, Haddad J, Freudenberg JM, Oommen DE, Hoffmann E, McCallum SW, Jacobson E. Assessing Colonic Exposure, Safety, and Clinical Activity of SRT2104, a Novel Oral SIRT1 Activator, in Patients with Mild to Moderate Ulcerative Colitis. Inflamm Bowel Dis. 2016 Mar;22(3):607-14. doi: 10.1097/MIB.0000000000000597. PMID 26595549
- See also: Results for study 115951 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115951?search=study&search_terms=115951#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115951 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register